CLINICAL TRIAL: NCT04091724
Title: Perioperative EEG-Monitoring and Emergence Delirium in Children: a Prospective Observational Study
Brief Title: Perioperative EEG-Monitoring and Emergence Delirium in Children
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua Zheng, Principal Investigator, Huazhong University of Science and Technology
Other Study IDs: TJMZK201901
Record Dates: First submitted 2019-09-10; First posted 2019-09-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium is determined by PAED score
- No delirium is determined by PAED score

SUMMARY:
Emergence delirium is a significant problem, particularly in children. However the incidence, preventative strategies, and management of emergence delirium remain unclear. Multichannel electroencephalogram is a recognized tool for identifying neurophysiologic states during anesthesia, sleep, and arousal. The aim of the current study is to evaluate the mechanisms and predictors of emergence delirium in children under 16 years scheduled for elective surgery using electroencephalogram. The "Pediatric Anesthesia Emergence Delirium Scores (PAED Score)" (Sikich et al. 2004) is used to screen for the occurrence of emergence delirium in the post anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

1. male or female children aged under 16 years
2. planned elective surgery
3. informed consent by parents or legal guardians

Exclusion Criteria:

1. history of neurological or psychiatric disease
2. delayed development
3. inability of the parents or legal guardians to speak or read Chinese
4. participation in another prospective interventional clinical study during this study

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children for elective surgery aged under 16 years
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence delirium | Recovery from anesthetic until discharge of the child from the Post-Anesthesia Care Unit, an average of 1 hour
  The Delirium is measured by the Pediatric Anesthesia Emergence Delirium Scores (PAED Score) (Sikich et al. 2004).The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity. A peak PAED value ≥ 10 is considered emergence delirium.

SECONDARY OUTCOMES:
Relative power of each brain waves | from stay at the preoperative holding room to discharge of the child from the Post-Anesthesia Care Unit, , an average of 3 hours
  Electroencephalogram data were acquired using a 32-channel electroencephalogram recording system (Brain Products, Germany). A 5 min, baseline, eyes-closed recording was conducted at the preoperative holding room when the child was at rest. Recording of electroencephalogram was commenced before the start of anesthetic induction and was stopped before discharge of the child from the Post-Anesthesia Care Unit. We defied delta (1 to 3 Hz), theta (4 to 7 Hz), alpha (8 to 12 Hz), and beta (13 to 40 Hz) frequency bands. And then, the relative power of each frequency bands to the total power of the sum is calculated.
Preoperative anxiety of children | baseline (At the preoperative holding room)
  Preoperative anxiety is evaluated using the preoperative modified Yale Preoperative Anxiety Scale (m-YPAS) score (Kain et al. 1997). The modified Yale Preoperative Anxiety Scale (m-YPAS) consists of 5 items (activity, vocalizations, emotional expressivity, state of apparent arousal, and use of parent). Children's behavior is rated from 1 to 4 or 1 to 6 (depending on the item), with higher numbers indicating the highest severity within that item. Each score is calculated by dividing each item rating by the highest possible rating (i.e., 6 for the "vocalizations" item and 4 for all other items), adding all the produced values, dividing by 5, and multiplying by 100. This calculation produces a score ranging from 23.33 to 100, with higher values indicating higher anxiety.
Compliance of the children during induction | Procedure (At the beginning of the Induction)
  Measured by Induction compliance checklist (Kain et al. 1998).
Blood pressure | During the operation, an average of 1 hour
  Systolic and diastolic blood pressures are assessed.
Heart rate | During the operation, an average of 1 hour
Body temperature | During the operation, an average of 1 hour
Duration of anesthesia | During the anesthesia, an average of 1 hour
Type of surgery | During the operation
Duration of surgery | During the operation, an average of 1 hour
Number of Participants with adverse events | Recovery from anesthetic until discharge of the child from the Post-Anesthesia Care Unit, , an average of 1 hour
  Adverse events such as vomiting, cough, breath holding, laryngospasm, and oxygen desaturation are recorded
The level of consciousness | Recovery from anesthetic until discharge of the child from the Post-Anesthesia Care Unit, an average of 1 hour
  The level of consciousness is measured by Richmond Agitation Sedation Scale score (Kerson et al. 2016). The Richmond Agitation and Sedation Scale (RASS) is a 10-point scale, with four levels of anxiety or agitation, one level denoting a calm and alert state, and 5 levels of sedation.
Postoperative pain: FLACC- Scale | Recovery from anesthetic until discharge of the child from the Post-Anesthesia Care Unit, an average of 1 hour
  Postoperative pain is measured by the FLACC- Scale (Merkel et al. 1997). The Face, Legs, Activity, Cry, Consolability (FLACC ) scale is a measurement used to assess pain for children or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Severity of emergence Delirium | Recovery from anesthetic until discharge of the child from the Post-Anesthesia Care Unit, an average of 1 hour
  The Delirium is measured by the Pediatric Anesthesia Emergence Delirium Scores (PAED Score) (Sikich et al. 2004).The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity. A peak PAED value ≥ 10 is considered emergence delirium.
Duration of emergence Delirium | Recovery from anesthetic until discharge of the child from the Post-Anesthesia Care Unit, an average of 1 hour
  The Delirium is measured by the Pediatric Anesthesia Emergence Delirium Scores (PAED Score) (Sikich et al. 2004).The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity. A peak PAED value ≥ 10 is considered emergence delirium.
Post-Anesthesia Care Unit (PACU) stay time | During the stay in the Post-Anesthesia Care Unit, an average of 1 hour
  When patients become calm and meet a modified Aldrete score (Aldrete et al. 1995) ≥ 9, they are discharged and the duration of the PACU stay is recorded as the PACU stay time.
Incidence of behavioral problem | Up to 30 postoperative days
  The behavioral problem is measured by a modified Version of the Posthospital Behavior Questionnaire (PHBQ) (Stargatt et al. 2006)
Number of Participants with postoperative organ complications | Participants will be followed for the duration of hospital stay, an average of 5 days.
Hospital length of stay | Participants will be followed for the duration of hospital stay, an average of 5 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kain ZN, Mayes LC, Wang SM, Caramico LA, Hofstadter MB. Parental presence during induction of anesthesia versus sedative premedication: which intervention is more effective? Anesthesiology. 1998 Nov;89(5):1147-56; discussion 9A-10A. doi: 10.1097/00000542-199811000-00015. PMID 9822003
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Stargatt R, Davidson AJ, Huang GH, Czarnecki C, Gibson MA, Stewart SA, Jamsen K. A cohort study of the incidence and risk factors for negative behavior changes in children after general anesthesia. Paediatr Anaesth. 2006 Aug;16(8):846-59. doi: 10.1111/j.1460-9592.2006.01869.x. PMID 16884468
- [Background] Kerson AG, DeMaria R, Mauer E, Joyce C, Gerber LM, Greenwald BM, Silver G, Traube C. Validity of the Richmond Agitation-Sedation Scale (RASS) in critically ill children. J Intensive Care. 2016 Oct 26;4:65. doi: 10.1186/s40560-016-0189-5. eCollection 2016. PMID 27800163